CLINICAL TRIAL: NCT04168593
Title: Randomized Controlled Trial of the Use of Acupuncture and Cupping in Patients Awaiting Total Knee Arthroplasty (TKA) Due to Knee Osteoarthritis
Brief Title: Association of Acupuncture and Cupping in Advanced Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Acupuncture in KOA
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2019-11

CONDITIONS: Knee Osteoarthritis; Pain, Chronic
Keywords: Acupuncture; Cupping; Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Osteoarthritis; Pain | interventions — Acupuncture Therapy; Cupping Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A- Placebo (Sham Comparator): Sham Acupuncture and Sham Cupping
  Interventions: Procedure: Acupuncture
- B -Cupping (Active Comparator): Sham Acupuncture and Real Cupping
  Interventions: Procedure: Acupuncture
- C - Acupuncture (Active Comparator): Real Acupuncture and Sham Cupping
  Interventions: Procedure: Acupuncture
- D - Acupuncture + Cupping (Active Comparator): Real Acupuncture and Real Cupping
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — 20 min of Acupuncture section follow by 10 min of cupping around the knee
  Other Names: Cupping

SUMMARY:
Given the lack of studies in the literature associating the use of acupuncture and sliding suction cup in patients with advanced knee osteoarthritis, the objective of this study is to evaluate the benefits of this association in patients of the Institute of Orthopedics and Traumatology outpatient clinic of the University of São Paulo while awaiting surgical treatment of knee osteoarthritis as a method of pain relief, limb function improvement and quality of life.

DETAILED DESCRIPTION:
120 patients with indications for surgical knee treatment from IOT-HCFMUSP will be invited to participate in the project. Inclusion applications and those who agree to sign a free and informed consent form (IC) will be included.

During the period of inclusion of patients, will be clarified regarding the application and evaluation methods that will be used through consultation and initial medical evaluation. Then, the included patients are randomized into four existing groups:

Group A - Acupuncture Sham + Cupping Sham; Group B - Sham Acupuncture + Real Cupping; Group C - Real Acupuncture + Sham Cupping; Group D - Real Acupuncture + Real Cupping.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of knee osteoarthritis
* WOMAC-Pain greater than or equal to 15 points.

Exclusion Criteria:

* advanced degenerative central neuropathy (Parkinson's, Alzheimer's)
* diabetic peripheral neuropathy
* stroke sequela
* history of digestive bleeding
* chronic renal failure
* renal failure
* heart failure
* fibromyalgia
* rheumatoid arthritis
* SLE
* severe depression
* psychiatric disorders
* concomitance with hip arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chin Lin, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- USaoPauloGH, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
these data are totally confidencial and unique to this protocol

REFERENCES:
- [Background] Kraus VB, Blanco FJ, Englund M, Karsdal MA, Lohmander LS. Call for standardized definitions of osteoarthritis and risk stratification for clinical trials and clinical use. Osteoarthritis Cartilage. 2015 Aug;23(8):1233-41. doi: 10.1016/j.joca.2015.03.036. Epub 2015 Apr 9. PMID 25865392
- [Result] Corbett MS, Rice SJ, Madurasinghe V, Slack R, Fayter DA, Harden M, Sutton AJ, Macpherson H, Woolacott NF. Acupuncture and other physical treatments for the relief of pain due to osteoarthritis of the knee: network meta-analysis. Osteoarthritis Cartilage. 2013 Sep;21(9):1290-8. doi: 10.1016/j.joca.2013.05.007. PMID 23973143

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment by phone from a list of patients with advanced KOA who is waiting for a TKR. the inclusion criteria is applied.
Pre-assignment Details: by phone we applied the WOMAC-Pain and invite who have 15 points or more
Groups:
- A- Acupuncture Sham + Cupping Sham: Sham acupuncture: Placement of placebo "dagger" needles. The needle tip, when touching the patient's skin, retracts into itself without puncturing the skin. Application locations: LI11, SP9, SP10, LR8, GB34, ST34, Ex-LE5. Running time of 20 minutes.
  Sham cupping: after each acupuncture session (Sham or True), the respective needles were removed, and acrylic suction cups were placed over the region where the needles were, attached to a strip (micropore) without exerting any negative pressure or movement. Application time of 10 minutes.
- B -Sham Acupuncture + Real Cupping: Acupuncture 20 min of Acupuncture section follow by 10 min of cupping around the knee
- C - Real Acupuncture + Sham Cupping; D - Real Acupuncture + Real Cupping: 20 min of Acupuncture section follow by 10 min of cupping around the knee
Period: Overall Study
Arm/Group | A- Acupuncture Sham + Cupping Sham | B -Sham Acupuncture + Real Cupping | C - Real Acupuncture + Sham Cupping | D - Real Acupuncture + Real Cupping
Started | 30 | 30 | 30 | 30
Completed | 26 | 28 | 27 | 29
Not Completed | 4 | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- A- Placebo: Sham Acupuncture and Sham Cupping
  20 min of Acupuncture section using placebo needle follow by 10 min of cupping sham (no negative pressure) around the knee
- B -Cupping: Sham Acupuncture and Real Cupping
  20 min of Acupuncture section using placebo needle follow by 10 min of real cupping around the knee
- C - Acupuncture: Real Acupuncture and Sham Cupping
  20 min of Real Acupuncture section follow by 10 min of sham cupping around the knee
- D - Acupuncture + Cupping: Real Acupuncture and Real Cupping
  20 min of Real Acupuncture section follow by 10 min of real cupping around the knee
- Total: Total of all reporting groups
Arm/Group | A- Placebo | B -Cupping | C - Acupuncture | D - Acupuncture + Cupping | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Customized [Mean (Standard Deviation); unit: years]
  Age distribution | 66.1 (10.88) | 66.1 (10.86) | 68.1 (11.15) | 66.8 (8.09) | 66.8 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 23 | 25 | 92
  Male | 9 | 7 | 7 | 5 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 30 | 30 | 30 | 120
WOMAC-Pain [Mean (Standard Deviation); unit: units on a scale] — range 0-20, 0 correspond to a better condition, otherwise, 20 correspond to a worst condition of pain
  units on a scale | 16.83 (1.74) | 16.50 (1.38) | 16.40 (1.43) | 16.90 (1.75) | 16.66 (1.58)
VAS [Mean (Standard Deviation); unit: units on a scale] — range 0-100, 0 correspond to a better condition, otherwise 100 correspond to a worst condition of pain
  units on a scale | 84.03 (13.75) | 89.57 (11.81) | 82.83 (12.97) | 91.30 (11.43) | 89.92 (12.88)

OUTCOME MEASURES:

1. Primary Outcome: WOMAC - Pain
Description: Western Ontario and McMaster Universities Osteoarthritis Womac-Pain section. Score: 0 (no pain) to 20 (worse condition)
Time Frame: value collected at 5 week
Population: We used the concept of Intent to Treat (ITT) for statistical analysis purposes, that is, all recruited participants, even if they did not complete the proposed 10-session treatment, were included in the final analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group A: Sham Acupuncture + Sham Cupping
- Group B: Sham Acupuncture + Real Cupping
- Group C: Real Acupuncture + Sham Cupping
- Group D: Real Acupuncture + Real Cupping
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 30 | 30 | 30 | 30
units on a scale | 11.60 (4.17) | 11.30 (4.23) | 10.80 (4.64) | 9.83 (4.76)

2. Primary Outcome: VAS
Description: Intensity of pain 0-100 mm (0 corresponds to a better condition, otherwise, 100 correspond to a worst condition of pain)
Time Frame: Value collected at 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 30 | 30 | 30 | 30
units on a scale | 67.43 (23.09) | 61.57 (25.57) | 47.87 (27.23) | 47.43 (28.99)

3. Secondary Outcome: Analgesic Consumption
Description: number of pills per day For each group, those who had a reduction in the use of pain medications (analgesics and/or anti-inflammatory drugs) we described as Y (yes), and those who maintained or even increased the amount or simply did not return such information we described as N (no).
Time Frame: Number of Participants with reduction in the use of pain medications after protocol (at 5 week)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Number of Participants With Reduction in the Use of Pain Medications: During the study, the name of the drug in use was noted, as well as its dosage, before and after the protocol.
Arm/Group | Number of Participants With Reduction in the Use of Pain Medications | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 120 | 30 | 30 | 30 | 30
Participants | 72 | 12 | 18 | 19 | 23

ADVERSE EVENTS:
Time Frame: after 5 weeks from initial treatment
Description: no serious adverse event, only local hematoma
Groups:
- Group A: Sham + Sham
- Group B: Sham Acp + Real Cupping
- Group C: Real ACP + Sham Cupping
- Group D: Real + Real
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 1/30 | 2/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=30) | Group B (N=30) | Group C (N=30) | Group D (N=30)
hematoma (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04168593/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04168593/SAP_001.pdf
  • Informed Consent Form (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04168593/ICF_002.pdf